CLINICAL TRIAL: NCT03928743
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Bimekizumab in Subjects With Active Ankylosing Spondylitis
Brief Title: A Study to Evaluate the Efficacy and Safety of Bimekizumab in Subjects With Active Ankylosing Spondylitis
Acronym: BE MOBILE 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AS0011; 2017-003065-95 (EudraCT Number)
Record Dates: First submitted 2019-04-23; First posted 2019-04-26 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing spondylitis; AS; Bimekizumab; Axial spondyloarthritis
MeSH Terms: conditions — Spondylitis, Ankylosing; Axial Spondyloarthritis | interventions — bimekizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bimekizumab (Experimental): Subjects randomized to this arm will receive bimekizumab during the Double-Blind Treatment Period and the Maintenance Period.
  Interventions: Drug: Bimekizumab
- Placebo (Placebo Comparator): Subjects randomized to this arm will receive placebo during the Double-Blind Treatment Period and receive bimekizumab during the Maintenance Period.
  Interventions: Drug: Bimekizumab; Other: Placebo

INTERVENTIONS:
Drug: Bimekizumab — Subjects will receive bimekizumab at pre-specified time-points.
  Other Names: BKZ; UCB4940
Other: Placebo — Subjects will receive placebo at pre-specified time-points during the Double-Blind Treatment Period.
  Other Names: PBO
  Arms: Placebo

SUMMARY:
The purpose of the study is to demonstrate the efficacy, safety and tolerability of bimekizumab administered subcutaneously (sc) compared to placebo in the treatment of subjects with active ankylosing spondylitis (AS).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients at least 18 years of age
* Subject has ankylosing spondylitis (AS) as per the Modified New York (mNY) criteria with documented radiologic evidence, and at least 3 months of symptoms with age at symptom onset less than 45 years
* Subjects has moderate-to-severe active disease defined by Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) >=4 AND spinal pain >=4 on a 0 to 10 Numeric Rating Scale
* Subjects had to have either failed to respond to 2 different nonsteroidal anti-inflammatory drugs (NSAIDs) given at the maximum tolerated dose for a total of 4 weeks or have a history of intolerance to or a contraindication to NSAID therapy
* Patients who have taken a tumor necrosis factor alpha (TNFα) inhibitor must have experienced an inadequate response or intolerance to treatment given at an approved dose for at least 12 weeks
* Patients currently taking NSAIDs, cyclooxygenase 2 (COX-2) inhibitors, analgesics, corticosteroids, methotrexate (MTX), leflunomide (LEF), sulfasalazine (SSZ), hydroxychloroquine (HCQ) AND/OR apremilast can be allowed if they fulfill specific requirements prior to study entry

Exclusion Criteria:

* Total ankylosis of the spine
* Treatment with more than 1 TNFα inhibitor and/or more than 2 additional non-TNFα biological response modifiers, or any interleukin (IL)-17 biological response modifier at any time are excluded
* Active infection or history of recent serious infections
* Viral hepatitis B or C or human immunodeficiency virus (HIV) infection
* Any live (includes attenuated) vaccination within the 8 weeks prior to entering the study or TB (Bacillus Calmette-Guerin) vaccination within 1 year prior entering the study
* Known tuberculosis (TB) infection, at high risk of acquiring TB infection, or current or history of nontuberculous mycobacterium (NTMB) infection
* Subject has any active malignancy or history of malignancy within 5 years prior to the Screening Visit EXCEPT treated and considered cured cutaneous squamous or basal cell carcinoma or in situ cervical cancer
* Diagnosis of inflammatory conditions other than AxSpA, eg, rheumatoid arthritis. Patients with a diagnosis of Crohn's disease, ulcerative colitis, or other inflammatory bowel disease (IBD) are allowed as long as they have no active symptomatic disease when entering the study.
* Presence of active suicidal ideation, or moderately severe major depression or severe major depression
* Female patients who are breastfeeding, pregnant, or planning to become pregnant during the study
* Subject has a history of chronic alcohol or drug abuse within 6 months prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2022-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (83):
- United States (14):
  - As0011 50131, Mesa, Arizona
  - As0011 50052, Phoenix, Arizona
  - As0011 50058, Phoenix, Arizona
  - As0011 50062, Sun City, Arizona
  - As0011 50060, Upland, California
  - As0011 50056, Sarasota, Florida
  - As0011 50015, Hagerstown, Maryland
  - As0011 50016, St Louis, Missouri
  - As0011 50054, Oklahoma City, Oklahoma
  - As0011 50020, Duncansville, Pennsylvania
  - As0011 50001, Jackson, Tennessee
  - As0011 50012, Memphis, Tennessee
  - As0011 50057, Dallas, Texas
  - As0011 50036, Mesquite, Texas
- Belgium (3):
  - As0011 40004, Brussels
  - As0011 40003, Genk
  - As0011 40001, Ghent
- Bulgaria (4):
  - As0011 40006, Plovdiv
  - As0011 40007, Plovdiv
  - As0011 40005, Sofia
  - As0011 40008, Sofia
- China (9):
  - As0011 20040, Beijing
  - As0011 20021, Chengdu
  - As0011 20019, Guangzhou
  - As0011 20034, Hefei
  - As0011 20024, Nanjing
  - As0011 20018, Shanghai
  - As0011 20020, Shanghai
  - As0011 20026, Shanghai
  - As0011 20025, Wenzhou
- Czechia (8):
  - As0011 40011, Brno
  - As0011 40009, Pardubice
  - As0011 40013, Prague
  - As0011 40014, Prague
  - As0011 40015, Prague
  - As0011 40016, Prague
  - As0011 40010, Uherské Hradiště
  - As0011 40012, Zlín
- France (2):
  - As0011 40018, Boulogne-Billancourt
  - As0011 40022, Limoges
- Germany (7):
  - As0011 40025, Berlin
  - As0011 40028, Berlin
  - As0011 40029, Hamburg
  - As0011 40024, Hanover
  - As0011 40027, Herne
  - As0011 40078, Leipzig
  - As0011 40026, Ratingen
- Hungary (4):
  - As0011 40032, Debrecen
  - As0011 40031, Szeged
  - As0011 40033, Székesfehérvár
  - As0011 40080, Szombathely
- Japan (11):
  - As0011 20030, Chūōku
  - As0011 20047, Himeji-shi
  - As0011 20045, Kita-gun
  - As0011 20065, Kitakyushu
  - As0011 20037, Osaka
  - As0011 20084, Saga
  - As0011 20048, Saitama
  - As0011 20031, Sapporo
  - As0011 20042, Sasebo
  - As0011 20032, Suita
  - As0011 20035, Tokyo
- As0011 40034, Amsterdam, Netherlands
- Poland (8):
  - As0011 40038, Elblag
  - As0011 40042, Krakow
  - As0011 40037, Lublin
  - As0011 40044, Poznan
  - As0011 40040, Torun
  - As0011 40041, Warsaw
  - As0011 40039, Wroclaw
  - As0011 40043, Wroclaw
- Spain (5):
  - As0011 40045, A Coruña
  - As0011 40046, Córdoba
  - As0011 40047, Madrid
  - As0011 40048, Santiago de Compostela
  - As0011 40049, Seville
- Turkey (Türkiye) (3):
  - As0011 40052, Ankara
  - As0011 40053, Ankara
  - As0011 40050, Istanbul
- United Kingdom (4):
  - As0011 40057, Edinburgh
  - As0011 40056, Leeds
  - As0011 40054, London
  - As0011 40055, Norwich

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org

REFERENCES:
- [Result] van der Heijde D, Deodhar A, Baraliakos X, Brown MA, Dobashi H, Dougados M, Elewaut D, Ellis AM, Fleurinck C, Gaffney K, Gensler LS, Haroon N, Magrey M, Maksymowych WP, Marten A, Massow U, Oortgiesen M, Poddubnyy D, Rudwaleit M, Shepherd-Smith J, Tomita T, Van den Bosch F, Vaux T, Xu H. Efficacy and safety of bimekizumab in axial spondyloarthritis: results of two parallel phase 3 randomised controlled trials. Ann Rheum Dis. 2023 Apr;82(4):515-526. doi: 10.1136/ard-2022-223595. Epub 2023 Jan 17. PMID 36649967
- [Result] Navarro-Compan V, Ramiro S, Deodhar A, Mease PJ, Rudwaleit M, de la Loge C, Fleurinck C, Taieb V, Morup MF, Massow U, Kay J, Magrey M. Association of clinical response criteria and disease activity levels with axial spondyloarthritis core domains: results from two phase 3 randomised studies, BE MOBILE 1 and 2. RMD Open. 2024 Apr 10;10(2):e004040. doi: 10.1136/rmdopen-2023-004040. PMID 38599650
- [Result] Dubreuil M, Navarro-Compan V, Boonen A, Gaffney K, Gensler LS, de la Loge C, Vaux T, Fleurinck C, Massow U, Taieb V, Morup MF, Deodhar A, Rudwaleit M. Improved physical functioning, sleep, work productivity and overall health-related quality of life with bimekizumab in patients with axial spondyloarthritis: results from two phase 3 studies. RMD Open. 2024 Jun 4;10(2):e004202. doi: 10.1136/rmdopen-2024-004202. PMID 38834351
- [Result] Ramiro S, Poddubnyy D, Mease PJ, Lopez-Medina C, Kim M, Massow U, Taieb V, Kragstrup TW, McGonagle D. Sustained resolution of enthesitis and peripheral arthritis over 104 weeks with bimekizumab in axial spondyloarthritis. RMD Open. 2025 Oct 22;11(4):e005969. doi: 10.1136/rmdopen-2025-005969. PMID 41125403
- [Derived] Marzo-Ortega H, Navarro-Compan V, Dubreuil M, Mease PJ, Magrey M, Rudwaleit M, D'Agostino MA, Gaffney K, Kay J, de la Loge C, Massow U, Taieb V, Vaux T, Deodhar A. Sustained improvements in spinal pain, morning stiffness, fatigue, sleep, physical function and overall health-related quality of life with bimekizumab in patients with axial spondyloarthritis: 2-year results from two phase 3 studies. RMD Open. 2025 Nov 28;11(4):e006013. doi: 10.1136/rmdopen-2025-006013. PMID 41314667
- [Derived] Mease PJ, Gensler LS, Orbai AM, Warren RB, Bajracharya R, Ink B, Marten A, Massow U, Shende V, Manente M, Peterson L, White K, Landewe R, Poddubnyy D. Long-term safety of bimekizumab in adult patients with axial spondyloarthritis or psoriatic arthritis: pooled results from integrated phase IIb/III clinical studies. RMD Open. 2025 Apr 6;11(2):e005026. doi: 10.1136/rmdopen-2024-005026. PMID 40194794
- [Derived] Navarro-Compan V, Rudwaleit M, Dubreuil M, Magrey M, Marzo-Ortega H, Mease PJ, Walsh JA, Dougados M, de la Loge C, Fleurinck C, Massow U, Vaux T, Taieb V, Deodhar A. Improved Pain, Morning Stiffness, and Fatigue With Bimekizumab in Axial Spondyloarthritis: Results From the Phase III BE MOBILE Studies. J Rheumatol. 2025 Jan 1;52(1):23-32. doi: 10.3899/jrheum.2024-0223. PMID 39406403
- [Derived] Cella D, de la Loge C, Fofana F, Guo S, Ellis A, Fleurinck C, Massow U, Dougados M, Navarro-Compan V, Walsh JA. The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) scale in patients with axial spondyloarthritis: psychometric properties and clinically meaningful thresholds for interpretation. J Patient Rep Outcomes. 2024 Aug 12;8(1):92. doi: 10.1186/s41687-024-00769-x. PMID 39133438
- [Derived] Baraliakos X, Deodhar A, van der Heijde D, Magrey M, Maksymowych WP, Tomita T, Xu H, Massow U, Fleurinck C, Ellis AM, Vaux T, Shepherd-Smith J, Marten A, Gensler LS. Bimekizumab treatment in patients with active axial spondyloarthritis: 52-week efficacy and safety from the randomised parallel phase 3 BE MOBILE 1 and BE MOBILE 2 studies. Ann Rheum Dis. 2024 Jan 11;83(2):199-213. doi: 10.1136/ard-2023-224803. PMID 37793792

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in April 2019 and concluded in August 2022.
Pre-assignment Details: The Participant Flow refers to the Randomized Set.
Groups:
- Placebo (up to Week 16): Participants received placebo matched to bimekizumab 160 milligrams (mg) every 4 weeks (Q4W) subcutaneously until Week 16.
- Bimekizumab 160 mg Q4W (up to Week 16): Participants received bimekizumab 160 mg Q4W subcutaneously until Week 16.
- Bimekizumab 160 mg Q4W (Week 16 up to Week 52): At the end of the 16-week Double-Blind Treatment Period, study participants receiving placebo were re-allocated to bimekizumab treatment at Week 16. All Participants received bimekizumab 160 mg Q4W subcutaneously from Week 16 until Week 48.
Period: Double-Blind Treatment Period:Weeks 1-16
Arm/Group | Placebo (up to Week 16) | Bimekizumab 160 mg Q4W (up to Week 16) | Bimekizumab 160 mg Q4W (Week 16 up to Week 52)
Started | 111 | 221 | 0
Completed | 109 | 213 | 0
Not Completed | 2 | 8 | 0
Not completed — Due To COVID-19 Pandemic and Site Restrictions | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Adverse Event, serious non-fatal | 0 | 1 | 0
Period: Maintenance Period: Weeks 16-52
Arm/Group | Placebo (up to Week 16) | Bimekizumab 160 mg Q4W (up to Week 16) | Bimekizumab 160 mg Q4W (Week 16 up to Week 52)
Started | 0 | 0 | 319 (Placebo=109 + BXZ=210 3 participants Completed the 16-Week Double-Blind Period but did not enter the Maintenance Period because of the below reason: Adverse event: 1 Withdrawal by study participants: 2)
Completed | 0 | 0 | 298
Not Completed | 0 | 0 | 21
Not completed — PI Decision Due To Non-Compliance and COVID 19 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 9
Not completed — Adverse event, serious non-fatal | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set which consisted of all randomized study participants who received at least one dose of the investigational medicinal product (IMP).
Groups:
- Placebo (up to Week 16): Participants received placebo matched to bimekizumab 160 mg Q4W subcutaneously until Week 16.
- Total: Total of all reporting groups
Arm/Group | Placebo (up to Week 16) | Bimekizumab 160 mg Q4W (up to Week 16) | Total
Number analyzed (Participants) | 111 | 221 | 332
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 109 | 212 | 321
  >=65 years | 2 | 9 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (12.6) | 41.0 (12.1) | 40.4 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 61 | 92
  Male | 80 | 160 | 240
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 20 | 37 | 57
  Black | 1 | 0 | 1
  White | 90 | 177 | 267
  Other/Mixed | 0 | 3 | 3
  Missing | 0 | 4 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 110 | 218 | 328
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Assessment of SpondyloArthritis International Society 40% Response Criteria (ASAS40) Response at Week 16
Description: ASAS40 response was defined as relative improvements of at least 40% and absolute improvement of at least 2 units on a 0 to 10 Numeric Rating Scale (NRS), where 0 is "not active" and 10 is "very active" in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PGADA) assessed disease activity on a scale of 0 [not active] to 10 [very active], higher score=more disease activity, Pain assessment on a scale of 0 [no pain] to 10 [most severe pain], higher score=more severity, Function (Bath Ankylosing Spondylitis Functional Index (BASFI)) assessed participant's level of ability on a scale of 0 [easy] to 10 [impossible], Inflammation (morning stiffness intensity and duration, mean of Q5 and Q6 of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) defined as 6 item questionnaire: measured disease activity on a scale of 0 [none] to 10 [severe], higher score=more disease activity) and no worsening at all in the remaining domain.
Time Frame: Week 16
Population: The Randomized Set consisted of all randomized study participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (up to Week 16) | Bimekizumab 160 mg Q4W (up to Week 16)
Number analyzed (Participants) | 111 | 221
percentage of participants | 22.5 | 44.8
Statistical Analysis 1: Comparison: Placebo (up to Week 16) vs Bimekizumab 160 mg Q4W (up to Week 16); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.88, 95% CI 2-sided [1.71 to 4.87]

2. Secondary Outcome: Percentage of Participants With Assessment of SpondyloArthritis International Society 40% Response Criteria (ASAS40) Response in TNFα Inhibitor-naïve Participants at Week 16
Description: ASAS40 response was defined as relative improvements of at least 40% and absolute improvement of at least 2 units on a 0 to 10 NRS, where 0 is "not active" and 10 is "very active" in at least 3 of the 4 domains: PGADA assessed disease activity on a scale of 0 [not active] to 10 [very active], higher score=more disease activity, Pain assessment on a scale of 0 [no pain] to 10 [most severe pain], higher score=more severity, Function (BASFI) assessed participant's level of ability on a scale of 0 [easy] to 10 [impossible], Inflammation (morning stiffness intensity and duration, mean of Q5 and Q6 of BASDAI defined as 6 item questionnaire: measured disease activity on a scale of 0 [none] to 10 [severe], higher score=more disease activity) and no worsening at all in the remaining domain.
Time Frame: Week 16
Population: The Randomized Set consisted of all randomized study participants. Here, Number of Participants Analyzed signifies those who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (up to Week 16) | Bimekizumab 160 mg Q4W (up to Week 16)
Number analyzed (Participants) | 94 | 184
percentage of participants | 23.4 | 45.7
Statistical Analysis 1: Comparison: Placebo (up to Week 16) vs Bimekizumab 160 mg Q4W (up to Week 16); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.80, 95% CI 2-sided [1.59 to 4.93]

3. Secondary Outcome: Percentage of Participants With Assessment of SpondyloArthritis International Society 20% Response Criteria (ASAS20) Response at Week 16
Description: ASAS20 response was defined as relative improvements of at least 20% and absolute improvement of at least 1 unit on a 0 to 10 NRS, where 0 is "not active" and 10 is "very active" in at least 3 of the 4 domains: PGADA assessed disease activity on a scale of 0 [not active] to 10 [very active], higher score=more disease activity, Pain assessment on a scale of 0 [no pain] to 10 [most severe pain], higher score=more severity, Function (BASFI) assessed participant's level of ability on a scale of 0 [easy] to 10 [impossible], Inflammation (morning stiffness intensity and duration, mean of Q5 and Q6 of BASDAI defined as 6 item questionnaire: measured disease activity on a scale of 0 [none] to 10 [severe], higher score=more disease activity) and no worsening at all in the remaining domain.
Time Frame: Week 16
Population: The Randomized Set consisted of all randomized study participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (up to Week 16) | Bimekizumab 160 mg Q4W (up to Week 16)
Number analyzed (Participants) | 111 | 221
percentage of participants | 43.2 | 66.1
Statistical Analysis 1: Comparison: Placebo (up to Week 16) vs Bimekizumab 160 mg Q4W (up to Week 16); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.66, 95% CI 2-sided [1.65 to 4.28]

4. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Total Score at Week 16
Description: BASDAI is a validated self-reported instrument, which consisted of 6 questions to measure the disease activity of ankylosing spondylitis (AS) from the participant's perspective. It measured the severity of fatigue, spinal and peripheral joint pain and swelling, enthesitis, and morning stiffness (both severity and duration). Each question was rated using a numerical rating scale from 0 (none) to 10 (very severe), higher score=high disease activity. The BASDAI score was calculated by computing the mean of questions 5 and 6 and adding it to the sum of questions 1 to 4. This score was then divided by 5. The total BASDAI score was ranged from 0=none to 10= very severe, where higher score indicated high disease activity. A negative value indicated improvement and a positive value indicated worsening.
Time Frame: Baseline, Week 16
Population: The Randomized Set consisted of all randomized study participants.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo (up to Week 16) | Bimekizumab 160 mg Q4W (up to Week 16)
Number analyzed (Participants) | 111 | 221
scores on a scale | -1.70 (0.21) | -2.74 (0.17)
Statistical Analysis 1: Comparison: Placebo (up to Week 16) vs Bimekizumab 160 mg Q4W (up to Week 16); Test type: Superiority; p < 0.001, Regression, Logistic; LS Mean difference = -1.04, 95% CI 2-sided [-1.48 to -0.59]

5. Secondary Outcome: Percentage of Participants With Assessment of SpondyloArthritis International Society (ASAS) Partial Remission (PR) at Week 16
Description: The Assessment of SpondyloArthritis International Society partial remission was defined as a score of less than or equal to (<=) 2 units (on a scale of 0-10, where 0=no disease activity and 10=high disease activity) in each of the 4 domains. These 4 domains included: PGADA assessed disease activity on a scale of 0 [not active] to 10 [very active], higher score=more disease activity, Pain assessment on a scale of 0 [no pain] to 10 [most severe pain], higher score=more severity, Function (BASFI) assessed participant's level of ability on a scale of 0 [easy] to 10 [impossible], Inflammation (morning stiffness intensity and duration, mean of Q5 and Q6 of BASDAI defined as 6 item questionnaire: measured disease activity on a scale of 0 [none] to 10 [severe], higher score=more disease activity).
Time Frame: Week 16
Population: The Randomized Set consisted of all randomized study participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (up to Week 16) | Bimekizumab 160 mg Q4W (up to Week 16)
Number analyzed (Participants) | 111 | 221
percentage of participants | 7.2 | 24.0
Statistical Analysis 1: Comparison: Placebo (up to Week 16) vs Bimekizumab 160 mg Q4W (up to Week 16); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.26, 95% CI 2-sided [1.93 to 9.39]

6. Secondary Outcome: Percentage of Participants With Ankylosing Spondylitis Disease Activity Score Major Improvement (ASDAS-MI) at Week 16
Description: ASDAS-MI is achieved when there is a reduction (improvement) of greater than or equal to (>=) 2.0 in the Ankylosing Spondylitis Disease Activity Score (ASDAS) relative to Baseline. ASDAS is calculated as the sum of the following components: 1) 0.121 × Total back pain (Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Q2 result), 2) 0.058 × Duration of morning stiffness (BASDAI Q6 result), 3) 0.110 × Patient's Global Assessment of Disease Activity (PGADA), 4) 0.073 × Peripheral pain/swelling (BASDAI Q3 result), 5) 0.579 × (natural logarithm of the C-reactive protein (CRP) [mg/L] + 1). Total back pain, PGADA, duration of morning stiffness, peripheral pain/swelling and fatigue are all assessed on a numerical scale (0 [no disease activity] to 10 [high disease activity] units). High ASDAS scores mean worse disease. If a participant achieves the ASDAS-MI it indicates a major improvement of their disease.
Time Frame: Week 16
Population: The Randomized Set consisted of all randomized study participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (up to Week 16) | Bimekizumab 160 mg Q4W (up to Week 16)
Number analyzed (Participants) | 111 | 221
percentage of participants | 5.4 | 25.8
Statistical Analysis 1: Comparison: Placebo (up to Week 16) vs Bimekizumab 160 mg Q4W (up to Week 16); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6.47, 95% CI 2-sided [2.67 to 15.65]

7. Secondary Outcome: Percentage of Participants With Assessment of SpondyloArthritis International Society (ASAS) 5/6 Response at Week 16
Description: The Assessment of SpondyloArthritis International Society (ASAS) 5/6 response is defined as achieving at least 20% improvement in 5 of 6 domains: PGADA assessed disease activity on a scale of 0 [not active] to 10 [very active], higher score=more disease activity, Pain assessment on a scale of 0 [no pain] to 10 [most severe pain], higher score=more severity), Function (BASFI) assessed participant's level of ability on a scale of 0 [easy] to 10 [impossible], Inflammation (morning stiffness intensity and duration, mean of Q5 and Q6 of BASDAI defined as 6 item questionnaire: measured disease activity on a scale of 0 [none] to 10 [severe], higher score=more disease activity), spinal mobility (lateral spinal flexion) and high sensitivity C-reactive protein (hs-CRP)].
Time Frame: Week 16
Population: The Randomized Set consisted of all randomized study participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (up to Week 16) | Bimekizumab 160 mg Q4W (up to Week 16)
Number analyzed (Participants) | 111 | 221
percentage of participants | 18.9 | 49.3
Statistical Analysis 1: Comparison: Placebo (up to Week 16) vs Bimekizumab 160 mg Q4W (up to Week 16); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.65, 4.65% CI 2-sided [2.51 to 7.57]

8. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 16
Description: The Bath Ankylosing Spondylitis Functional Index (BASFI) assesses physical function in comprising 10 items relating to activities during the past week. Each item ranged from 0 ('Easy') to 10 ('Impossible'). The BASFI is the mean of the 10 scores such that the total score ranges from 0 to 10, with lower scores indicating better physical function. A negative value in BASFI change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Time Frame: Baseline, Week 16
Population: The Randomized Set consisted of all randomized study participants.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo (up to Week 16) | Bimekizumab 160 mg Q4W (up to Week 16)
Number analyzed (Participants) | 111 | 221
scores on a scale | -0.95 (0.20) | -2.00 (0.16)
Statistical Analysis 1: Comparison: Placebo (up to Week 16) vs Bimekizumab 160 mg Q4W (up to Week 16); Test type: Superiority; p < 0.001, Regression, Logistic; LS Mean difference = -1.05, 95% CI 2-sided [-1.48 to -0.63]

9. Secondary Outcome: Change From Baseline in Nocturnal Spinal Pain Score Numeric Rating Scale (NRS) at Week 16
Description: Nocturnal spinal pain experienced by ankylosing spondylitis (AS) participants is measured by one question: pain in the spine at night due to AS?. When responding, the participant is to consider the average amount of pain in the preceding week. It is assessed on a numerical scale of 0 (no pain) to 10 (most severe pain) units. A lower score indicates less pain and a negative change represents an improvement.
Time Frame: Baseline, Week 16
Population: The Randomized Set consisted of all randomized study participants.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo (up to Week 16) | Bimekizumab 160 mg Q4W (up to Week 16)
Number analyzed (Participants) | 111 | 221
scores on a scale | -1.68 (0.25) | -3.16 (0.20)
Statistical Analysis 1: Comparison: Placebo (up to Week 16) vs Bimekizumab 160 mg Q4W (up to Week 16); Test type: Superiority; p < 0.001, Regression, Logistic; LS Mean difference = -1.48, 95% CI 2-sided [-2.00 to -0.96]

10. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Quality of Life (ASQoL) Total Score at Week 16
Description: The Ankylosing Spondylitis Quality of Life (ASQoL), a validated disease-specific 18-item questionnaire, has been developed specifically for measuring health-related quality of life (HRQoL) in participants with ankylosing spondylitis and has shown to be responsive in axial spondyloarthritis (axSpA). Each statement on the ASQoL is given a score of 1=Yes or 0=No. A score of "1" was given where the item was affirmed, indicating adverse quality of life. All item scores were summed to generate the total score ranging from 0 to 18 with a higher score indicating worse health-related quality of life. A negative change from baseline represents an improvement.
Time Frame: Baseline, Week 16
Population: The Randomized Set consisted of all randomized study participants.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo (up to Week 16) | Bimekizumab 160 mg Q4W (up to Week 16)
Number analyzed (Participants) | 111 | 221
scores on a scale | -3.07 (0.41) | -4.59 (0.32)
Statistical Analysis 1: Comparison: Placebo (up to Week 16) vs Bimekizumab 160 mg Q4W (up to Week 16); Test type: Superiority; p < 0.001, Regression, Logistic; LS Mean difference = -1.52, 95% CI 2-sided [-2.36 to -0.68]

11. Secondary Outcome: Change From Baseline in the Short Form 36-Item Health Survey (SF-36) Physical Component Summary (PCS) Score at Week 16
Description: SF-36 is a 36-item HRQoL instrument with recall period of 4 weeks. Items are grouped into 8 domains: Physical Functioning (10 items), Role Physical (4 items), Bodily Pain (2 items), General Health (5 items), Vitality (4 items), Social Functioning (2 items), Role Emotional (3 items), Mental Health (5 items) and 1 item for Health Transition during last year. PCS and Mental Component Summary (MCS) scores are calculated from 8 domains (excluding Health Transition item). Each of SF-36 derived raw scores range from 0 to 100; higher score = better function. PCS score is calculated from 8 domain scores. It is standardized score ranging from 7.3 to 70.1, with a mean of 50 and SD of 10 in general US population, higher values = better function, and positive change reflects improvement. A PCS score mean below 47 indicates impaired physical functioning. Individual respondent's score that falls outside T-score range of 45 to 55 are outside average general US population range.
Time Frame: Baseline, Week 16
Population: The Randomized Set consisted of all randomized study participants.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo (up to Week 16) | Bimekizumab 160 mg Q4W (up to Week 16)
Number analyzed (Participants) | 111 | 221
T-score | 5.17 (0.82) | 8.54 (0.67)
Statistical Analysis 1: Comparison: Placebo (up to Week 16) vs Bimekizumab 160 mg Q4W (up to Week 16); Test type: Superiority; p < 0.001, Regression, Logistic; LS Mean difference = 3.38, 95% CI 2-sided [1.67 to 5.09]

12. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Metrology Index (BASMI) at Week 16
Description: The Bath Ankylosing Spondylitis Disease Metrology Index characterizes the spinal mobility of participants with axial Spondyloarthritis (SpA) and Ankylosing Spondylitis. It is a disease-specific measure consisting of 5 clinical measures to reflect participant axial status: cervical rotation; tragus to wall distance; lateral lumbar flexion; lumbar flexion (modified Schober test); intermalleolar distance. According to the linear definition of the BASMI a score of 0 to 10 was calculated for each item based on the measurement. The mean of the 5 scores provides the total BASMI score (ranging from 0 to 10). The higher the BASMI score, the more severe the participant's limitation of movement due to their axial SpA. A negative value in BASMI change from Baseline indicates an improvement from Baseline. The higher the negative value, the better the improvement.
Time Frame: Baseline, Week 16
Population: The Randomized Set consisted of all randomized study participants.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo (up to Week 16) | Bimekizumab 160 mg Q4W (up to Week 16)
Number analyzed (Participants) | 111 | 221
scores on a scale | -0.17 (0.09) | -0.45 (0.07)
Statistical Analysis 1: Comparison: Placebo (up to Week 16) vs Bimekizumab 160 mg Q4W (up to Week 16); Test type: Superiority; p = 0.006, Regression, Logistic; LS Mean difference = -0.28, 95% CI 2-sided [-0.47 to -0.08]

13. Secondary Outcome: Change From Baseline in the Maastricht Ankylosing Spondylitis Enthesitis (MASES) Index in the Subgroup of Participants With Enthesitis at Baseline at Week 16
Description: The Maastricht Ankylosing Spondylitis Enthesitis is an index that measures the severity (ie, intensity and extent) of enthesitis through the assessment of 13 entheses (bilateral costochondral 1, costochondral 7, anterior superior iliac spine, posterior iliac spine, iliac crest and proximal insertion of the Achilles tendon sites, and the fifth lumbar vertebral body spinous process), each scored as 0 or 1 and then summed for a possible score of 0 to 13. A higher score reflects higher severity and a negative change represents an improvement.
Time Frame: Baseline, Week 16
Population: Subset of study participants in Randomized Set with enthesitis at Baseline.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo (up to Week 16) | Bimekizumab 160 mg Q4W (up to Week 16)
Number analyzed (Participants) | 67 | 132
scores on a scale | -1.04 (0.33) | -2.12 (0.26)
Statistical Analysis 1: Comparison: Placebo (up to Week 16) vs Bimekizumab 160 mg Q4W (up to Week 16); Test type: Superiority; p = 0.003, Regression, Logistic; LS Mean difference = -1.08, 95% CI 2-sided [-1.79 to -0.38]

14. Secondary Outcome: Percentage of Participants With Enthesitis-free State at Week 16 Based on the Maastricht Ankylosing Spondylitis Enthesitis Index in the Subgroup of Participants With Enthesitis at Baseline
Description: The Maastricht Ankylosing Spondylitis Enthesitis is an index that measures the severity (ie, intensity and extent) of enthesitis through the assessment of 13 entheses (bilateral costochondral 1, costochondral 7, anterior superior iliac spine, posterior iliac spine, iliac crest and proximal insertion of the Achilles tendon sites, and the fifth lumbar vertebral body spinous process) each scored as 0 or 1 and then summed for a possible score of 0 to 13. Enthesitis free state is defined as having a MASES score of 0. A higher score reflects higher severity and a negative change represents an improvement.
Time Frame: Baseline, Week 16
Population: Subset of study participants in Randomized Set with enthesitis at Baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (up to Week 16) | Bimekizumab 160 mg Q4W (up to Week 16)
Number analyzed (Participants) | 67 | 132
percentage of participants | 32.8 | 51.5
Statistical Analysis 1: Comparison: Placebo (up to Week 16) vs Bimekizumab 160 mg Q4W (up to Week 16); Test type: Superiority; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 2.47, 95% CI 2-sided [1.30 to 4.68]

15. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) During the Study
Description: TEAEs are defined as those AEs that have a start date on or following the first dose of study treatment through the final dose of study treatment + 140 days (covering the 20-week Safety follow up (SFU) period). TEAEs were analyzed and have been reported for Double Blind Treatment Period (Safety set),Maintenance Period (MP) (Maintenance Set) and Overall Period (Safety set) which includes all participants who received BKZ 60 mg Q4W during the study.
Time Frame: From Baseline (Day 1) until Safety-Follow-Up (up to Week 68)
Population: The Safety Set consisted of all randomized study participants who received at least one dose of the IMP.
Measure: Number; unit: percentage of participants
Groups:
- Double Blind Treatment Period (up to Week 16): Placebo: Participants received placebo matched to bimekizumab 160 mg Q4W subcutaneously until Week 16.
- Double Blind Treatment Period (up to Week 16): Bimekizumab 160 mg Q4W: Participants received bimekizumab 160 mg Q4W subcutaneously until Week 16.
- Maintenance Period (Week 16 up to Week 52): Bimekizumab 160 mg Q4W: At the end of the 16-week Double-Blind Treatment Period, study participants receiving placebo were re-allocated to bimekizumab treatment at Week 16. All Participants received bimekizumab 160 mg Q4W subcutaneously from Week 16 until Week 48.
- Overall Period (up to Week 48 + 20 Weeks SFU): Bimekizumab 160 mg Q4W: Participants who received bimekizumab 160 mg Q4W subcutaneously from Day 1 and participants who switched from placebo arm at Week 16 to receive bimekizumab 160 mg Q4W subcutaneously were included in this group.
Arm/Group | Double Blind Treatment Period (up to Week 16): Placebo | Double Blind Treatment Period (up to Week 16): Bimekizumab 160 mg Q4W | Maintenance Period (Week 16 up to Week 52): Bimekizumab 160 mg Q4W | Overall Period (up to Week 48 + 20 Weeks SFU): Bimekizumab 160 mg Q4W
Number analyzed (Participants) | 111 | 221 | 319 | 330
percentage of participants | 43.2 | 54.3 | 68.3 | 75.8

16. Secondary Outcome: Percentage of Participants With Treatment-emergent Serious Adverse Events (SAEs) During the Study
Description: A serious adverse event (SAE) is any untoward medical occurrence that at any dose resulted in 1) Death, 2) Life-threatening (Life-threatening does not include a reaction that might have caused death had it occurred in a more severe form.), 3) Significant or persistent disability/incapacity, 4) Congenital anomaly/birth defect (including that occurring in a fetus), 5) Important medical event that, based upon appropriate medical judgment, may jeopardize the participant or participant may require medical or surgical intervention to prevent 1 of the other outcomes listed in the definition of serious (Important medical events may include, but are not limited to, potential Hy's Law [see allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.)
Time Frame: From Baseline (Day 1) until Safety-Follow-Up (up to Week 68)
Population: The Safety Set consisted of all randomized study participants who received at least one dose of the IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Double Blind Treatment Period (up to Week 16): Placebo | Double Blind Treatment Period (up to Week 16): Bimekizumab 160 mg Q4W | Maintenance Period (Week 16 up to Week 52): Bimekizumab 160 mg Q4W | Overall Period (up to Week 48 + 20 Weeks SFU): Bimekizumab 160 mg Q4W
Number analyzed (Participants) | 111 | 221 | 319 | 330
percentage of participants | 0.9 | 2.3 | 4.7 | 6.1

17. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) Leading to Withdrawal From Investigational Medicinal Product (IMP) During the Study
Description: TEAEs are defined as those AEs that have a start date on or following the first dose of study treatment through the final dose of study treatment + 140 days (covering the 20-week SFU period).
Time Frame: From Baseline (Day 1) until Safety-Follow-Up (up to Week 68)
Population: The Safety Set consisted of all randomized study participants who received at least one dose of the IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Double Blind Treatment Period (up to Week 16): Placebo | Double Blind Treatment Period (up to Week 16): Bimekizumab 160 mg Q4W | Maintenance Period (Week 16 up to Week 52): Bimekizumab 160 mg Q4W | Overall Period (up to Week 48 + 20 Weeks SFU): Bimekizumab 160 mg Q4W
Number analyzed (Participants) | 111 | 221 | 319 | 330
percentage of participants | 0 | 3.2 | 2.8 | 4.8

ADVERSE EVENTS:
Time Frame: From Baseline (Day 1) until Safety-Follow-Up (up to Week 68)
Description: As pre-specified in SAP, Maintenance Period (MP) included adverse events of Safety follow up period for participants who did not enter the open label extension or discontinued early in MP. TEAEs were analyzed and have been reported for Double Blind Treatment Period (Safety set),MP (Maintenance Set) and Overall Period (Safety set) which includes all participants who received BKZ 60 mg Q4W during the study.
Arm/Group | Double Blind Treatment Period (up to Week 16): Placebo | Double Blind Treatment Period (up to Week 16): Bimekizumab 160 mg Q4W | Maintenance Period (Week 16 up to Week 52): Bimekizumab 160 mg Q4W | Overall Period (up to Week 48 + 20 Weeks SFU): Bimekizumab 160 mg Q4W
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/221 | 0/319 | 0/330
Serious Adverse Events (participants affected / at risk) | 1/111 | 5/221 | 15/319 | 20/330
Other Adverse Events (participants affected / at risk) | 16/111 | 43/221 | 64/319 | 95/330
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Blind Treatment Period (up to Week 16): Placebo (N=111) | Double Blind Treatment Period (up to Week 16): Bimekizumab 160 mg Q4W (N=221) | Maintenance Period (Week 16 up to Week 52): Bimekizumab 160 mg Q4W (N=319) | Overall Period (up to Week 48 + 20 Weeks SFU): Bimekizumab 160 mg Q4W (N=330)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatitis A (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Superficial spreading melanoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinoplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Blind Treatment Period (up to Week 16): Placebo (N=111) | Double Blind Treatment Period (up to Week 16): Bimekizumab 160 mg Q4W (N=221) | Maintenance Period (Week 16 up to Week 52): Bimekizumab 160 mg Q4W (N=319) | Overall Period (up to Week 48 + 20 Weeks SFU): Bimekizumab 160 mg Q4W (N=330)
Nasopharyngitis (Infections and infestations) | 4 (4) | 17 (21) | 17 (18) | 30 (39)
Upper respiratory tract infection (Infections and infestations) | 8 (11) | 6 (6) | 16 (17) | 21 (23)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 7 (7) | 12 (15) | 18 (22)
Oral Candidiasis (Infections and infestations) | 0 (0) | 10 (11) | 12 (14) | 20 (25)
Headache (Nervous system disorders) | 5 (5) | 9 (10) | 11 (13) | 18 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT03928743/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT03928743/SAP_001.pdf